CLINICAL TRIAL: NCT02364414
Title: The Accuracy of Direct Digital Intra-oral Scanning Measurements Compared to Measurements on Study Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering General Hospital NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Rdb394 v6.1
Record Dates: First submitted 2015-01-28; First posted 2015-02-18 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Orthodontics; Study Models; Intra-oral Scanning; Measurements; Digital; Three Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Other): Orthodontic patients, aged 11-18 who fulfill the inclusion/exclusion criteria and provide written informed consent to participate will undergo intra-oral scan. This will be repeated 2 weeks later.
  Interventions: Device: 3Shape TRIOS (R)

INTERVENTIONS:
Device: 3Shape TRIOS (R) — Direct intra-oral scan of teeth and dentition

SUMMARY:
The purpose of this study is to compare the accuracy of measurements derived from a commercially available direct intra-oral scanning system with those taken from plaster study models, and to compare cost implications of both systems.

The investigators will test the hypotheses:

* There is no systematic difference between measurements taken from the Trios scanner and study models.
* There is no difference in the cost of producing digital models.

DETAILED DESCRIPTION:
Plaster study models produced from moulds of the teeth are a standard component of orthodontic records. They are fundamental to diagnosis and treatment planning, evaluation of treatment progress and results as well as record keeping. (Santoro et al., 2003) Plaster models must be retained for a minimum of 11 years for a medico legal reasons. This leads to problems of storage in terms of space and cost, in addition to the risk of damage because of the brittle nature of the models. These problems therefore highlight the need for an alternative method for producing and storing study models. This study aims to compare the accuracy of measurements derived from a new commercially available direct intra-oral (inside of the mouth) scanning system (3Shape TRIOS (R)) with those taken from plaster study models, and to compare cost implications of both systems. We will use the results to conclude whether direct intra¬oral scanning can replace traditional plaster models produced from moulds of the teeth.

ELIGIBILITY:
Inclusion Criteria:

* Age range 11 years old to 18 years old.
* Orthodontic patients with a range of malocclusions.
* Dentition without abnormal morphology.
* Adult/permanent dentition from the first molar to first molar in both arches.

Exclusion Criteria:

* Patients under 11 years old and over 18 years old.
* Carious teeth or teeth with significantly altered anatomy.
* Periodontal disease with significant gingival swelling.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measurement of tooth widths, arch lengths, overjet, overbite, crown heights and labio lingual widths | Within six weeks of initial intervention
  All dental study models, and 3D scans will have all the above measurements carried out. There are 22 patients and each will have had study models made and these will be measured twice on two separate occasions, and all scans measured twice.
  The measurements will be compared and analysed to see if the 3D scans accurately represent the tooth sizes and measurements that have been carried out on the dental study models (gold standard).

SECONDARY OUTCOMES:
Cost | within 6 months of initial intervention
  To determine the difference in cost between the two systems

CONTACTS AND LOCATIONS:
Overall Officials: Julian O'Neill, BDS FFDRCS MOrth, Principal Investigator — Kettering General Hospital NHS Foundation Trust
Locations (1):
- Kettering General Hospital NHS Foundation Trust, Kettering, Northamptonshire, United Kingdom

REFERENCES:
- [Background] Santoro M, Galkin S, Teredesai M, Nicolay OF, Cangialosi TJ. Comparison of measurements made on digital and plaster models. Am J Orthod Dentofacial Orthop. 2003 Jul;124(1):101-5. doi: 10.1016/s0889-5406(03)00152-5. PMID 12867904
- [Background] Han UK, Vig KW, Weintraub JA, Vig PS, Kowalski CJ. Consistency of orthodontic treatment decisions relative to diagnostic records. Am J Orthod Dentofacial Orthop. 1991 Sep;100(3):212-9. doi: 10.1016/0889-5406(91)70058-5. PMID 1877545
- [Background] Rheude B, Sadowsky PL, Ferriera A, Jacobson A. An evaluation of the use of digital study models in orthodontic diagnosis and treatment planning. Angle Orthod. 2005 May;75(3):300-4. doi: 10.1043/0003-3219(2005)75[300:AEOTUO]2.0.CO;2. PMID 15898364
- [Background] Fleming PS, Marinho V, Johal A. Orthodontic measurements on digital study models compared with plaster models: a systematic review. Orthod Craniofac Res. 2011 Feb;14(1):1-16. doi: 10.1111/j.1601-6343.2010.01503.x. Epub 2010 Nov 22. PMID 21205164
- [Background] Cuperus AM, Harms MC, Rangel FA, Bronkhorst EM, Schols JG, Breuning KH. Dental models made with an intraoral scanner: a validation study. Am J Orthod Dentofacial Orthop. 2012 Sep;142(3):308-13. doi: 10.1016/j.ajodo.2012.03.031. PMID 22920696
- [Background] Bell A, Ayoub AF, Siebert P. Assessment of the accuracy of a three-dimensional imaging system for archiving dental study models. J Orthod. 2003 Sep;30(3):219-23. doi: 10.1093/ortho/30.3.219. PMID 14530419
- [Background] Lee SP, Delong R, Hodges JS, Hayashi K, Lee JB. Predicting first molar width using virtual models of dental arches. Clin Anat. 2008 Jan;21(1):27-32. doi: 10.1002/ca.20580. PMID 18092365
- [Background] Machen DE. Legal aspects of orthodontic practice: risk management concepts. The diagnostic dilemma. Am J Orthod Dentofacial Orthop. 1991 Apr;99(4):381-2. doi: 10.1016/s0889-5406(05)81419-2. No abstract available. PMID 2008899
- [Background] Tomassetti JJ, Taloumis LJ, Denny JM, Fischer JR Jr. A comparison of 3 computerized Bolton tooth-size analyses with a commonly used method. Angle Orthod. 2001 Oct;71(5):351-7. doi: 10.1043/0003-3219(2001)0712.0.CO;2. PMID 11605868
- [Background] Zilberman O, Huggare JA, Parikakis KA. Evaluation of the validity of tooth size and arch width measurements using conventional and three-dimensional virtual orthodontic models. Angle Orthod. 2003 Jun;73(3):301-6. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 12828439
- [Background] Quimby ML, Vig KW, Rashid RG, Firestone AR. The accuracy and reliability of measurements made on computer-based digital models. Angle Orthod. 2004 Jun;74(3):298-303. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15264638
- [Background] Keim RG, Gottlieb EL, Nelson AH, Vogels DS 3rd. 2008 JCO study of orthodontic diagnosis and treatment procedures, part 1: results and trends. J Clin Orthod. 2008 Nov;42(11):625-40. No abstract available. PMID 19075377
- [Background] Mayers M, Firestone AR, Rashid R, Vig KW. Comparison of peer assessment rating (PAR) index scores of plaster and computer-based digital models. Am J Orthod Dentofacial Orthop. 2005 Oct;128(4):431-4. doi: 10.1016/j.ajodo.2004.04.035. PMID 16214623
- [Background] Pani SC, Hedge AM. Impressions in cleft lip and palate--a novel two stage technique. J Clin Pediatr Dent. 2008 Winter;33(2):93-6. PMID 19358372
- [Background] Sousa MV, Vasconcelos EC, Janson G, Garib D, Pinzan A. Accuracy and reproducibility of 3-dimensional digital model measurements. Am J Orthod Dentofacial Orthop. 2012 Aug;142(2):269-73. doi: 10.1016/j.ajodo.2011.12.028. PMID 22858338
- [Background] Kachalia PR, Geissberger MJ. Dentistry a la carte: in-office CAD/CAM technology. J Calif Dent Assoc. 2010 May;38(5):323-30. PMID 20572526
- [Background] Meyer BJ, Mormann WH, Lutz F. [Optimization of the powder application in the Cerec method with environment-friendly propellant systems]. Schweiz Monatsschr Zahnmed. 1990;100(12):1462-8. German. PMID 2277979